CLINICAL TRIAL: NCT00000762
Title: A Placebo-Controlled, Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Envelope Proteins of HIV-1 gp160 and gp120 in Children >= 1 Month Old With Asymptomatic HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry); MicroGeneSys Inc (nka Protein Sciences Corporation) (Unknown)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 218; 11195 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV Envelope Protein gp160; HIV Envelope Protein gp120; AIDS Vaccines; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections | interventions — VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: rgp120/HIV-1MN
Biological: rgp120/HIV-1 SF-2
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
To determine the safety and immunogenicity of gp160 (MicroGeneSys), rgp120/HIV-1MN (Genentech), and rgp120/HIV-1SF2 (BIOCINE) and their adjuvants in HIV-infected children 1 month to 18 years of age.

The initiation of this immunotherapy trial will provide multiple benefits by assessing in asymptomatic HIV-infected children a therapy currently being tested in their adult counterparts, in the hope of forestalling the progression of HIV immunosuppression and clinical disease.

DETAILED DESCRIPTION:
The initiation of this immunotherapy trial will provide multiple benefits by assessing in asymptomatic HIV-infected children a therapy currently being tested in their adult counterparts, in the hope of forestalling the progression of HIV immunosuppression and clinical disease.

Patients are randomized to receive one of three vaccines (9 patients/vaccine) or the adjuvant placebos (3 patients/vaccine). The vaccines will be studied at both low and high doses. When three of four patients at the low dose of a vaccine have received two immunizations without evidence of dose-limiting toxicity, dose escalation to the higher dose of that vaccine is initiated in subsequent patient cohorts, provided all low dose arms are filled. A total of six immunizations are given, at 0, 4, 8, 12, 16, and 24 weeks. Patients are followed for 24 weeks after the last immunization.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication: Recommended:

* PCP prophylaxis.

Patients must have:

* Documented asymptomatic HIV infection.
* CD4+ count as follows:
* 1-11 months of age must have > 2000 cells/mm3 and >= 30 percent of the total lymphocytes; 12-23 months must have > 1000 cells/mm3 and >= 20 percent of the total lymphocytes; 24 months-6 years must have > 750 cells/mm3 and >= 20 percent of the total lymphocytes; and 7 years and older must have > 500 cells/mm3 and >= 20 percent of the total lymphocytes.

NOTE:

* Patients who received zidovudine for 3 consecutive months immediately prior to study entry may receive only high doses of vaccine.

Exclusion Criteria

Co-existing Condition:

Patients with the following condition are excluded:

* Any serious acute infection.

Concurrent Medication:

Excluded:

* Anticipated steroid therapy of > 6 weeks duration.

Excluded within the past 2 years:

* More than one serious proven bacterial infection such as sepsis, pneumonia, meningitis, bone or joint infection, abscess of an internal organ or body cavity (other than otitis media or superficial skin or mucosal abscesses) caused by Haemophilus, Streptococcus, Pneumococcus, or other pyogenic bacteria.

Prior Medication:

Excluded:

* Antiretroviral therapy or immunomodulators (e.g., IVIG) within 1 month prior to study entry (NOTE: AZT is allowed within 1 month prior to study entry if patient is entering a high-dose arm).
* Uninterrupted steroid therapy of > 6 weeks duration.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72
Dates: Study Completion 1996-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lambert JS, Study Chair; Katz S, Study Chair
Locations (34):
- United States (33):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Childrens Hosp. LA - Dept. of Ped., Div. of Clinical Immunology & Allergy, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - San Francisco Gen. Hosp., San Francisco, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Connecticut Health Ctr., Dept. of Ped., Farmington, Connecticut
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Cook County Hosp., Chicago, Illinois
  - Univ. of Illinois College of Medicine at Chicago, Dept. of Peds., Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - UMDNJ - Robert Wood Johnson, New Brunswick, New Jersey
  - NJ Med. School CRS, Newark, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey, Paterson, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - North Shore-Long Island Jewish Health System, Dept. of Peds., Great Neck, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - Texas Children's Hosp. CRS, Houston, Texas
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Lambert JS, McNamara J, Katz S, Fenton T, Nichols J, Roberts NJ. Safety and immunogenicity of recombinant envelope HIV vaccines in asymptomatic HIV-infected children. Natl Conf Hum Retroviruses Relat Infect (1st). 1993 Dec 12-16:72
- [Background] Lambert JS, et al. Safety and immunogenicity of recombinant envelope HIV vaccines in asymptomatic HIV infected children. Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:151
- [Background] Lambert JS, McNamara J, Katz SL, Fenton T, Kang M, VanCott TC, Livingston R, Hawkins E, Moye J Jr, Borkowsky W, Johnson D, Yogev R, Duliege AM, Francis D, Gershon A, Wara D, Martin N, Levin M, McSherry G, Smith G. Safety and immunogenicity of HIV recombinant envelope vaccines in HIV-infected infants and children. National Institutes of Health-sponsored Pediatric AIDS Clinical Trials Group (ACTG-218). J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Dec 15;19(5):451-61. doi: 10.1097/00042560-199812150-00003. PMID 9859958
- [Background] Lambert JS, McNamara J, Katz S, Livingston R, Moye J. Safety and immunogenicity of HIV recombinant envelope vaccines in HIV-infected infants and children. Pediatric AIDS Clinical Trials Group Study ACTG 218. American Pediatric Association and Society for Pediatric Research annual meeting; 1996 May 6-10; Washington, D.C. Pediatr AIDS HIV Infect. 1996 Aug;7(4):279 (unnumbered abstract)
- [Result] Lambert JS. HIV vaccines in infants and children. Paediatr Drugs. 2005;7(5):267-76. doi: 10.2165/00148581-200507050-00001. PMID 16220994